CLINICAL TRIAL: NCT05272085
Title: Comparison of the Efficacy of Ultrasound-Guided Lavage and Subacromial Bursa Injection in Calcific Tendinitis: A Prospective, Randomized, Double-Blind Study
Brief Title: Comparison of the Efficiency of Ultrasound-Guided Lavage and Subacromial Bursa Injection in Calcific Tendinitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Nuri Tugbay Yildiran, Principal Investigator, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IstanbulUC-NTugbayYildiran-01
Record Dates: First submitted 2022-02-20; First posted 2022-03-09 (Actual); Last update posted 2023-01-31 (Actual); Status verified 2023-01

CONDITIONS: Calcific Tendinitis; Calcific Tendinitis of Shoulder; Shoulder Pain
Keywords: Calcific tendinitis; Shoulder pain; Ultrasound-guided; Lavage; Barbotage; subacromial bursa injection
MeSH Terms: conditions — Rotator Cuff Tear Arthropathy; Shoulder Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ultrasound Guided Lavage Group (Active Comparator): The physical examination, pain scoring, functional scale, disability scale, special tests, direct radiography findings and ultrasonographic imaging findings of the patients in this group before the treatment and 1 month after the treatment will be evaluated and will be recorded. Size of calcific deposits and Gartner classification will be evaluated on direct radiography. Size, shape, acoustic shadowing, power doppler activity of calcific deposits and other bursitis, tendinitis, ruptures, effusion in the shoulder will be evaluated on ultrasonographic imaging.
  Patients in this group will be treated with ultrasound-guided lavage.
  Interventions: Procedure: Ultrasound Guided Lavage
- Ultrasound Guided Subacromial Bursa Injection Group (Active Comparator): The physical examination, pain scoring, functional scale, disability scale, special tests, direct radiography findings and ultrasonographic imaging findings of the patients in this group before the treatment and 1 month after the treatment will be evaluated and will be recorded. Size of calcific deposits and Gartner classification will be evaluated on direct radiography. Size, shape, acoustic shadowing, power doppler activity of calcific deposits and other bursitis, tendinitis, ruptures, effusion in the shoulder will be evaluated on ultrasonographic imaging.
  Patients in this group will be treated with ultrasound-guided subacromial bursa injection with corticosteroid and lidocaine.
  Interventions: Procedure: Ultrasound Guided Subacromial Bursa Injection

INTERVENTIONS:
Procedure: Ultrasound Guided Lavage — After local anesthesia of subcutaneous tissue, lavage will be performed under the guidance of ultrasound using an 18-gauge needle with injectors filled with 4 ml of saline. The needle will be advanced to the center of the calcific deposit. The injector will be kept as parallel to the ground as possible. The plunger of the injector will be pushed with a gently pressure and then released. Calcific deposits are expected to be filled into the syringe along with saline. It is predicted that the clear saline will gradually turn white and become cloudy due to the incoming calcific deposits. When the color of the liquid becomes cloudy, the syringe will be removed without moving the needle, and a new syringe containing 4 ml saline will be placed in its place. Thus, the aspirated calcific deposits will not be reinjected. The same process will be repeated with a new saline filled syringe. After the procedure, 2 ml dexamethasone and 3 ml lidocaine will be injected in subacromial bursa.
  Other Names: Ultrasound Guided Barbotage
  Arms: Ultrasound Guided Lavage Group
Procedure: Ultrasound Guided Subacromial Bursa Injection — 2 ml dexamethasone and 3 ml %2 lidocaine will be injected in the subacromial bursa using a 21-gauge needle under ultrasound guidance.
  Arms: Ultrasound Guided Subacromial Bursa Injection Group

SUMMARY:
It is aimed to compare in the early period the clinical and ultrasonographic findings in terms of the effectiveness of ultrasound-guided subacromial bursa injection with corticosteroid and ultrasound-guided lavage, which are the treatment options available in the literature for patients with calcific tendinitis who do not respond to conservative treatment.

DETAILED DESCRIPTION:
Calcific tendinitis is a disease that occurs with the precipitation of hydroxyapatite crystals on tendons and shoulder region is the most involved. In the shoulder region, calcific tendinitis can involve all rotator cuff tendons, most commonly the supraspinatus. It may progress with pain and functional limitation. The pain can increase with movement or can occur at rest and sleep. The prevalence of calcific tendinitis is between 2.7% and 20% in the general population. The most common age group is between 30 and 60. It can negatively affect the family and social life of the person and cause loss of workforce.

Especially in the treatment of patients with calcific tendinitis unresponsive to conservative treatment, ultrasound-guided corticosteroid injection in subacromial bursa and ultrasound-guided lavage are frequently used treatment options. However, there are very few studies in the literature comparing these two treatment methods as randomized controlled trials.

In this study, it is aimed to compare the effectiveness of ultrasound guided subacromial bursa injection and ultrasound guided lavage procedures on pain scores, functional scales, disability scales, direct radiography findings and ultrasonographic imaging findings.

ELIGIBILITY:
Inclusion Criteria:

* Cases diagnosed with calcific tendinitis who did not benefit from conservative treatment
* Cases with calcific deposits greater than 1 cm in direct radiography, ultrasonography, or magnetic resonance imaging
* Cases between the ages of 18-75 whose informed consent was obtained for participation in the study

Exclusion Criteria:

* Cases with radiculopathy ipsilateral to the affected shoulder
* Cases with active inflammatory arthropathy of the affected shoulder
* Cases with previous shoulder surgery
* Cases with a history of humeral head, scapula, and clavicle fractures
* Cases with neurological deficit affecting the upper extremity
* Cases with uncontrolled diabetes mellitus and uncontrolled hypertension, uncompensated congestive heart failure, chronic renal failure, chronic liver disease, tumor and/or vascular disease, inflammatory and/or infectious diseases, currently active psychiatric disease
* Cases with a history of subacromial bursa injection, calcific lavage or shoulder joint injection in the last 3 months
* Cases with a history of allergic reaction to the substance to be applied as local anesthetic
* Pregnancy or lactation
* Anticoagulant or antiagregant (antiplatelet) medication use that may interfere with the injection procedure.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2022-03-09 (Actual); Primary Completion 2022-08-30 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
Change of Range of Motion | Baseline, 1 month
  The change in a participant's range of motion degree as measured by a goniometer (Passive Range of Motion and Active Range of Motion) from baseline to 1 month.
Clinical improvement measured by change in Numeric Rating Scale | Baseline, 1 hour, 1 month
  A numerical rating scale (NRS) requires the patient to rate their pain on a defined scale. A patient selects a whole number (0-10 integers) that best reflects the intensity of his/her pain. The 11-point numeric scale ranges from '0' representing "no pain" to '10' representing "worst possible pain"
Clinical improvement measured by change in Constant Shoulder Score | Baseline, 1 month
  The constant shoulder score is a validated scale, measuring the shoulder function. It is an objective measurement independent of the shoulder pain. It is a 100-points scale composed of a number of individual parameters. The minimum score is 0, the maximum score is 100 points. The higher the score, the higher the quality of the function.
Clinical improvement measured by change in Quick Dash Score | Baseline, 1 month
  Individual's ability to complete tasks, absorb forces, and severity of symptoms are measured by a 11 item Quick Dash questionnaire. At least 10 of the 11 items must be completed for a score to be calculated and the scores range from 0 (no disability) to 100 (most severe disability).
Clinical improvement measured by change in Shoulder Disability Questionnaire | Baseline, 1 month
  This score measures the disability of the shoulder in daily life, work, social life.0 points indicate maximum well-being, 100 points indicate maximum disability
Change in Gartner Score of the Shoulder Calcifications on Direct Radiography | Baseline, 1 month
  Radiological classification of calcifying tendinitis
Change in ultrasound scoring system presented by Chiou | Baseline, 1 month
  This score includes size, shape (arc, fragmented, nodular, cystic), power doppler activity of calcific deposits.
Change in ultrasound classification system of calcific deposits presented by Farin | Baseline, 1 month
  This classification includes acoustic shadowing of calcific deposits (well-defined shadow, faint shadow and no shadow)

CONTACTS AND LOCATIONS:
Overall Officials: NURI TUGBAY YILDIRAN, Principal Investigator — Istanbul University - Cerrahpasa; DENIZ PALAMAR, Study Director — Istanbul University - Cerrahpasa; BILGE CAKIR, Study Chair — Istanbul University - Cerrahpasa
Locations (1):
- Istanbul University- Cerrahpaşa, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Louwerens JK, Sierevelt IN, van Hove RP, van den Bekerom MP, van Noort A. Prevalence of calcific deposits within the rotator cuff tendons in adults with and without subacromial pain syndrome: clinical and radiologic analysis of 1219 patients. J Shoulder Elbow Surg. 2015 Oct;24(10):1588-93. doi: 10.1016/j.jse.2015.02.024. Epub 2015 Apr 11. PMID 25870115
- [Background] Sansone V, Maiorano E, Galluzzo A, Pascale V. Calcific tendinopathy of the shoulder: clinical perspectives into the mechanisms, pathogenesis, and treatment. Orthop Res Rev. 2018 Oct 3;10:63-72. doi: 10.2147/ORR.S138225. eCollection 2018. PMID 30774461
- [Background] Sansone V, Consonni O, Maiorano E, Meroni R, Goddi A. Calcific tendinopathy of the rotator cuff: the correlation between pain and imaging features in symptomatic and asymptomatic female shoulders. Skeletal Radiol. 2016 Jan;45(1):49-55. doi: 10.1007/s00256-015-2240-3. Epub 2015 Aug 27. PMID 26306389
- [Background] Greis AC, Derrington SM, McAuliffe M. Evaluation and nonsurgical management of rotator cuff calcific tendinopathy. Orthop Clin North Am. 2015 Apr;46(2):293-302. doi: 10.1016/j.ocl.2014.11.011. Epub 2015 Jan 27. PMID 25771323
- [Background] de Witte PB, Selten JW, Navas A, Nagels J, Visser CP, Nelissen RG, Reijnierse M. Calcific tendinitis of the rotator cuff: a randomized controlled trial of ultrasound-guided needling and lavage versus subacromial corticosteroids. Am J Sports Med. 2013 Jul;41(7):1665-73. doi: 10.1177/0363546513487066. Epub 2013 May 21. PMID 23696211
- [Background] Chiou HJ, Chou YH, Wu JJ, Hsu CC, Huang DY, Chang CY. Evaluation of calcific tendonitis of the rotator cuff: role of color Doppler ultrasonography. J Ultrasound Med. 2002 Mar;21(3):289-95; quiz 296-7. doi: 10.7863/jum.2002.21.3.289. PMID 11883540
- [Background] Farin PU, Jaroma H. Sonographic findings of rotator cuff calcifications. J Ultrasound Med. 1995 Jan;14(1):7-14. doi: 10.7863/jum.1995.14.1.7. PMID 7707483
- [Background] Gartner J, Heyer A. [Calcific tendinitis of the shoulder]. Orthopade. 1995 Jun;24(3):284-302. German. PMID 7617385
- [Background] Zhang T, Duan Y, Chen J, Chen X. Efficacy of ultrasound-guided percutaneous lavage for rotator cuff calcific tendinopathy: A systematic review and meta-analysis. Medicine (Baltimore). 2019 May;98(21):e15552. doi: 10.1097/MD.0000000000015552. PMID 31124934
- [Background] Lee S.H. (2020) Calcific Tendinitis Intervention. In: Peng P., Finlayson R., Lee S., Bhatia A. (eds) Ultrasound for Interventional Pain Management. Springer, Cham. https://doi.org/10.1007/978-3-030-18371-4_26